CLINICAL TRIAL: NCT02025647
Title: An Open, Non-Randomized, Evaluation of Innerview™, an MHCDS Tool Used to Report Symptoms and Functioning Related to Common Mental Health Disorders in the Primary Care Setting
Brief Title: An Evaluation of Innerview™, a Web-based Tool to Support the Integration of Mental Health in the Primary Care Setting
Status: Completed | Type: Observational
Sponsor: Pearson/Clinical Assessment (Industry)
Responsible Party: Sponsor
Other Study IDs: IV-0022
Record Dates: First submitted 2013-12-22; First posted 2014-01-01 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Mental Health
Keywords: Mood disorders; Anxiety disorders; Eating concerns; Pain concerns; Alcohol abuse; Self harm; Mental health; Clinical Decision Support
MeSH Terms: conditions — Psychological Well-Being; Mood Disorders; Anxiety Disorders; Alcoholism; Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Innerview MHCDS: Innerview, Mental Health Clinical Decision Support tool

SUMMARY:
Innerview can address some of the challenges of integrating mental health and primary care by accurately and reliably collecting mental health evidence and activities directly from patients, and then organizing and automating that evidence and activity into reports for providers and care teams that support diagnosis, treatment planning and monitoring of the mental health issues within a practice population.

DETAILED DESCRIPTION:
To deliver integrated quality care, innovative strategies are needed to efficiently collect, understand, monitor and manage mental health evidence and its contribution to the primary care office visit. Computer applications can provide solutions to providers by helping their processes to be feasible, manageable, and sustainable. We hypothesize that by both providing patients the opportunity to reflect on their physical, emotional and behavioral symptoms and functioning, and giving providers accurate, reliable, current, symptom-based mental health evidence in an accessible organized format prior to the face-to-face visit, Innerview will enhance diagnostic and treatment processes from both a patient- and population-based perspective, as well as enhance communication between patient and provider.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria:

  * Provide signed and dated informed consent form
  * Be aged 18 or older
  * Be willing to comply with all study procedures and be available for the duration of the study
  * Be able to read English at an 8th grade level (as determined by physician)
  * Have internet access to email with a computer and/or tablet

Exclusion Criteria:

* Patients are excluded from study participation if they meet any of the following criteria:

  * Inability to provide consent due to guardianship issues
  * Currently experiencing psychotic symptoms (as determined by physician)
  * Anything that, in the opinion of the Investigator, would preclude the subject's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Innerview will be given universally / as indicated to 150 non-randomly selected subjects aged 18 and over seeking primary care in selected primary care study sites.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sloan Manning, MD, Principal Investigator — Novant Healthcare; Sherry Falsetti, PhD, Principal Investigator — University of Illinois at Chicago; Donald Nease, MD, Principal Investigator — University of Colorado, Denver; Peter J Knoblich, MD, Principal Investigator — Peter J. Knoblich MD; William Ervin, MD, Principal Investigator — Intermed, PA
Locations (5):
- United States (5):
  - Peter J. Knoblich MD, Roseville, California
  - University of Colorado, Denver, Colorado
  - University of Illinois, Rockford, Illinois
  - Intermed, PA, Portland, Maine
  - Novant Healthcare, Winston-Salem, North Carolina

REFERENCES:
- [Background] Katon W, Von Korff M, Lin E, Unutzer J, Simon G, Walker E, Ludman E, Bush T. Population-based care of depression: effective disease management strategies to decrease prevalence. Gen Hosp Psychiatry. 1997 May;19(3):169-78. doi: 10.1016/s0163-8343(97)00016-9. PMID 9218985
- [Background] Wang PS, Demler O, Olfson M, Pincus HA, Wells KB, Kessler RC. Changing profiles of service sectors used for mental health care in the United States. Am J Psychiatry. 2006 Jul;163(7):1187-98. doi: 10.1176/ajp.2006.163.7.1187. PMID 16816223
- See also: Mental Health: A Report of the Surgeon General — http://profiles.nlm.nih.gov/ps/retrieve/ResourceMetadata/NNBBHS
- See also: Prevalence of serious mental illness among U.S. adults by age, sex, and race — http://nimh.nih.gov/statistics/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is comprised of a series of 3 study sessions spanning a maximum participation period of 30-45 days. All subjects are intended to complete Study Session 1 and 2, spanning a duration of 24-48 hours. Those subjects who endorsed enough diagnostic symptoms to generate an Individualized Rating Scale will participate through Study Session 3.
Period: Overall Study
Arm/Group | Innerview MHCDS
Started | 139
Session 1 (Narrative Module) | 139
Immediate Retest (Rating Module: 5 Min) | 97 (27 did not generate IRS 15 technology issues or administered wrong session)
Session 2 (Narrative Module: 24-48 Hrs) | 117 (19 lost to follow up or technology issues 3 administered wrong session)
Session 3 (Rating Module: 30-45 Days) | 76 (27 did not generate IRS 36 lost to follow up)
Completed | 139
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 139
Age, Customized [Number; unit: participants]
  18-40 years | 46
  41-60 years | 38
  61+ years | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 50
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 15
  Hispanic | 5
  White | 117
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 139
Those with and w/o mental health concerns as identified by each investigator [Number; unit: participants]
  With Mental Health Concerns | 35
  Without Mental Health Concerns | 104

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of the Narrative Module
Description: Out of 139 subjects using Innerview for the first time, how many subjects approved their initial version of their narrative versus chose to start over?
Time Frame: Immediate
Measure: Number; unit: participants
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 139
participants | 139

2. Primary Outcome: Reliability of the Narrative Module
Description: What is the consistency of the diagnostic criteria generated by two administrations, 1 to 2 days apart?
Time Frame: 24-48 hours
Measure: Mean (Standard Deviation); unit: percentage of agreement
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 117
percentage of agreement | 94 (5)

3. Primary Outcome: Standard Error of Measure for the Individualized Rating Scale (Rating Module)
Description: What is the standard error of measurement (SEM) for test/retest symptom ratings on a 0 - 10 point scale
Time Frame: approximate 5 minutes between ratings
Measure: Number; unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 97
units on a scale | .9

4. Secondary Outcome: Provider Survey (Question 1)
Description: The information provided by Innerview is valuable in understanding and treating my patients.
  Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Administered Innerview session on at least 15 subjects
Population: This is an investigator survey meant to measure the usefullness, feasibility and acceptability of the tool. Therefore, this question was not asked of the subjects but of their providers. There were a total of 6 providers/investigators that enrolled 15 or more subjects.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 6
units on a scale | 4.5 [1 to 5]

5. Secondary Outcome: Provider Survey (Question 2)
Description: The information provided by Innerview was consistent with my previous observations of my patients.
  Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Administered Innerview session on at least 15 subjects
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 6
units on a scale | 4.3 [1 to 5]

6. Secondary Outcome: Provider Survey (Question 3)
Description: The information provided by Innerview was well organized in the reports. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Administered Innerview session on at least 15 subjects
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 6
units on a scale | 4.3 [1 to 5]

7. Secondary Outcome: Provider Survey (Question 4)
Description: The information provided by Innerview was well communicated in the reports. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Administered Innerview session on at least 15 subjects
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 6
units on a scale | 4.3 [1 to 5]

8. Secondary Outcome: Provider Survey (Question 5)
Description: In my opinion, the Innerview narrative process will help prepare patients for treatment.
  Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Administered Innerview session on at least 15 subjects
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 6
units on a scale | 3.5 [1 to 5]

9. Secondary Outcome: Provider Survey (Question 6)
Description: Innerview will help me better identify patients who suffer from a mental health concern.
  Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Administered Innerview session on at least 15 subjects
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 6
units on a scale | 3.7 [1 to 5]

10. Secondary Outcome: Provider Survey (Question 7)
Description: Innerview will function well within my current work flow Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Administered Innerview session on at least 15 subjects
Population: This is an investigator survey meant to measure the usefullness, feasibility and acceptability of the tool. Therefore, this question was not asked of the subjects but of their providers. There were a total of 6 providers/investigators that enrolled 15 or more subjects, one investigator did not respond to this item.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 6
units on a scale | 4.2 [1 to 5]

11. Secondary Outcome: Provider Survey (Question 8)
Description: My patients reacted positively to Innerview. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Administered Innerview session on at least 15 subjects
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 6
units on a scale | 4.2 [1 to 5]

12. Secondary Outcome: Provider Survey (Question 9)
Description: In my opinion, incorporating Innerview into my practice would require an acceptable amount of time and effort from myself and staff Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Administered Innerview session on at least 15 subjects
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 6
units on a scale | 3.2 [1 to 5]

13. Secondary Outcome: Provider Survey (Question 10)
Description: The benefits of Innerview will outweigh the effort to implement and operate it. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Administered Innerview session on at least 15 subjects
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 6
units on a scale | 3.5 [1 to 5]

14. Secondary Outcome: Provider Survey (Question 11)
Description: On average, how much extra time do you estimate that you spent with your patients evaluating and discussing the information collected through Innerview?
Time Frame: Administered Innerview session on at least 15 subjects
Population: as for outcome 4
Measure: Mean (Full Range); unit: minutes
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 6
minutes | 15 [3 to 30]

15. Secondary Outcome: Subject Survey (Question 1)
Description: I am satisfied with how I was able to tell my story. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 135
units on a scale | 4.03 (.73)

16. Secondary Outcome: Subject Survey (Question 2)
Description: Compared to other health care questionnaires I have taken, I would rate this system highly.
  Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 132
units on a scale | 3.89 (.78)

17. Secondary Outcome: Subject Survey (Question 3)
Description: The program was easy to use. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 132
units on a scale | 3.89 (.92)

18. Secondary Outcome: Subject Survey (Question 4)
Description: This tool will contribute positively to my health care. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 135
units on a scale | 4.39 (.61)

19. Secondary Outcome: Subject Survey (Question 5)
Description: The program included all of the symptoms I wanted to share with my doctor. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 126
units on a scale | 4.44 (.59)

20. Secondary Outcome: Subject Survey (Question 6)
Description: I was able to select words and phrases that I normally use to talk about my symptoms.
  Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 132
units on a scale | 4.25 (.72)

21. Secondary Outcome: Subject Survey (Question 7)
Description: Q7. I would encourage other doctors to use this system. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 115
units on a scale | 4.10 (.74)

22. Secondary Outcome: Subject Survey (Question 8)
Description: Telling my story helped me prepare for treatment. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 118
units on a scale | 3.81 (.82)

23. Secondary Outcome: Subject Survey (Question 9)
Description: The demonstration showed me how to use the system. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 128
units on a scale | 3.95 (.75)

24. Secondary Outcome: Subject Survey (Question 10)
Description: It took an acceptable amount of time to tell my story. Where 1 is strongly disagree 2 is disagree 3 is neutral 4 is agree 5 is strongly agree
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 133
units on a scale | 4.11 (.70)

25. Other Pre Specified Outcome: Completion Times
Description: On average, the number of minutes taken to complete both the narrative and rating modules?
Time Frame: Study Duration
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 97
minutes | 15.56 [9.49 to 23.11]

26. Post Hoc Outcome: Mental Health Prevalence Rates Comparison
Description: What is the percentage of subjects where the provider was unaware of any mental health concerns yet Innerview identified them as having hit a rule out or diagnostic consideration for a mental health disorder vs the US 12 Month Prevalence Rate?
  US 12 Month Prevalence Rate = 26.2% (http://www.ncbi.nlm.nih.gov/pubmed/15939839)
Time Frame: Study Duration
Population: 104 subjects had no known mental health concerns
Measure: Number; unit: percentage of subjects
Arm/Group | Innerview MHCDS
Number analyzed (Participants) | 104
percentage of subjects | 27

ADVERSE EVENTS:
Time Frame: Study duration
Arm/Group | Innerview MHCDS
Serious Adverse Events (participants affected / at risk) | 0/139
Other Adverse Events (participants affected / at risk) | 0/139

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No